CLINICAL TRIAL: NCT04758169
Title: Improving Nutrition, Health and Livelihoods Through Enhanced Homestead Food Production: A Strategy to Reduce Child Marriage in Bangladesh
Brief Title: Exploring Enhanced HFP to Reduce Child Marriage in Bangladesh
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Helen Keller International (Other)
Collaborators: International Development Research Centre, Canada (Other Government); Mount Saint Vincent University (Other)
Responsible Party: Principal Investigator, Asif Chowdhury, Head of Monitoring, Evaluation and Research, Helen Keller International
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 35923112020
Record Dates: First submitted 2021-02-10; First posted 2021-02-17 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Adolescent Behavior; Health Behavior; Marriage Age
Keywords: Homestead Food Production; Sexual and Reproductive Health; Dietary Diversity; Household Food Security
MeSH Terms: conditions — Adolescent Behavior; Health Behavior; Coitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Homestead Food Production (Experimental): Participant in this arm will receive the Helen Keller's EHFP model which involves homestead food production, nutrition and WASH education and gender transformative sessions (intervention group). Participants will also receive interventions related to parental awareness sessions, community awareness-raising activities, adolescent group sessions involving awareness on the benefit of delayed marriage and empowerment, SRH and basic life-skill trainings.
  Interventions: Other: Enhanced Homestead Food Production
- Control (Experimental): Participants in this arm will only receive parental awareness sessions, community awareness-raising activities, adolescent group sessions involving awareness on the benefit of delayed marriage and empowerment, SRH, and basic life-skill trainings. This particular arm will not receive any homestead food production intervention over the course of the implementation.
  Interventions: Other: Control

INTERVENTIONS:
Other: Enhanced Homestead Food Production — Enhanced Homestead Food Production program will provide increased production and consumption of nutrient rich foods, increased income of the households through the sale of surplus produce, and increased self-efficacy and decision making by adolescents due to increased knowledge and skills- resulting increased food security and nutrition and ultimately delay of child marriage.
  Arms: Enhanced Homestead Food Production
Other: Control — Control group will only receive parental awareness sessions, community awareness-raising activities, adolescent group sessions involving awareness on the benefit of delayed marriage and empowerment, SRH, and basic life-skill trainings.
  Arms: Control

SUMMARY:
Child marriage leads to pregnancy in adolescence, a root cause of both malnutrition and the intergenerational cycle of malnutrition. Two-thirds of Bangladeshi girls are married before 18 years, nearly half become pregnant before 19, and the rates of stunting and underweight are 26% and 36%, respectively. There are well-established risks of adolescent pregnancy for both mother (impaired growth and development due to nutrient reallocation for pregnancy and lactation), and infants (increased risk of low birth weight and small-for-gestational-age). Poor sexual and reproductive health (SRH), infant and young child feeding (IYCF), and water, sanitation, and hygiene (WASH) knowledge could impair the nutritional and health status of the whole family, sparking intergenerational issues.

The investigators propose to investigate the efficacy of a gender-transformative enhanced homestead food production (EHFP) program to prevent child marriage, and in turn, adolescent pregnancy-induced malnutrition among girls aged 13-15 years in a high-risk area for child marriage, Khulna Division, southern Bangladesh. The investigators will conduct a cluster-randomized controlled trial in which n=1200 girls in after-school Adolescent Clubs will participate in a 24-month program teaching women's empowerment through hands-on workshops. All participants (control and EHFP groups) will be exposed to SRH, WASH, and IYCF, while those in the EHFP group will also receive EFHP training and inputs intended to improve nutrient intake and provide an income source for the adolescent girls' family.

Investigators hypothesize that girls in the EHFP group will have lower rates of marriage and pregnancy, and improved food security, dietary diversity, nutritional status, IYCF, WASH, and SRH knowledge/practices.

DETAILED DESCRIPTION:
Introduction: Over the past 20 years, Bangladesh has heavily invested in improving the health and nutrition status of its adolescent population, however despite this investment, adolescents remain a vulnerable group. A recent large scale survey found that 26% of adolescents were stunted and 36% had low BMI(1). Nationally, 31% of married adolescent girls between the ages of 15 to 19 years were found to be underweight and another 13 percent were stunted (2). Adolescent women's sexual and reproductive health (SRH) knowledge is also a concern in Bangladesh, as unmarried adolescents have little access to SRH services (3). Adolescent health status is further exacerbated by high fertility rates with two-thirds of Bangladeshi women married before their eighteenth birthday while almost half of women are under 19 years at the time of their first pregnancy (4). Furthermore, data from the Bangladesh Integrated Households Survey 2017 reports that more than half of the children born to women under 15 were stunted while only 51% of married adolescents were using modern contraceptives (5). Statistics are worse in southern Bangladesh, particularly in Khulna Division, where the average age at first marriage is 15.5 years, with more than 8% experiencing birth intervals of less than 24 months and 32% of married adolescents age 15-19 years not using any form of contraceptive (5).

Adolescents are an important target group as they have the potential to contribute to society and earn income for their full adult life in addition to the intergenerational impact of undernourished teens having undernourished children, adversely impacting the health of future generations as well as long term human capital (6). Adolescents face risks as they move from adolescence to adulthood including poor nutritional status, inadequate (SRH) knowledge, insufficient education, early marriage, early pregnancy and social stigma (1,7). Lack of SRH has a direct impact on health and nutrition. For the past several decades, various organizations including the National Nutrition Services (NNS) in the Directorate General of Health Services (DGHS) under the Ministry of Health, Ministry of Women and Child Affairs (MoWCA); Non-Governmental Organizations; and Civil Society Organizations have undertaken initiatives to address issues related to ensuring the overall wellbeing of the adolescents. Such interventions have often been fragmented with limited scalability, sustainability and replicability. Since the improvement of adolescent nutrition in multifaceted, these efforts lacked a full-service delivery approach that would enable a comprehensive and systematic multisectoral engagement. Moreover, detailed evidence regarding the long-term effectiveness of such efforts in reaching their overarching goals is limited. The Ministry of Women and Children Affairs (MOWCA) has initiated the Adolescent Club Program of Bangladesh to mainstream SRH education through a club-based intervention to empower adolescents but which is limited to improving SRH knowledge(8).

In 2019, Helen Keller International in collaboration with the Mount Saint Vincent University, Canada (MSVU) initiated a three year research project in Debhata Sub-District of the Satkhira District in Khulna Division, funded by the International Research and Development Center (IDRC) Canada to increase production of diversified and nutrient-rich food, increase income generation from transferred assets, access to income, and access to improved knowledge and awareness on nutrition and adolescents along with essential nutrition actions and essential hygiene actions. SRH information is also included to improve outcomes including self-efficacy and agency to delay child marriage. These activities are underscored by a transformative approach to gender equality at the household and community level to improve intra-household communication and respect and intra-community equality and inclusion.

Objectives: To establish whether a gender transformative enhanced homestead food production (EHFP) model can improve household food security, diet, nutrition, income, and sexual and reproductive health outcomes to delay child marriage among Bangladeshi girls.

Specific objectives:

1. Test the effect of an integrated gender transformative Enhanced Homestead Food Production (EHFP) model on household food security
2. Assess the impact of household and community level interventions on adolescent dietary quality, nutritional status and prevalence of anemia.
3. Identify the threshold of income generated through EHFP that influences family decisions to delay child marriage.
4. Identify the determinants of adolescent empowerment and participation in household decision-making through EHFP.
5. Inform and contribute to evidence-based policy and decision making related to nutrition, health, income generation, SRH and delayed age of marriage.

Methodology: The investigators propose to investigate the efficacy of a gender-transformative Enhanced Homestead Food Production (EHFP) program to prevent child marriage, and in turn, adolescent pregnancy-induced malnutrition among girls aged 13-15 years in a high-risk area for child marriage, Khulna Division, southern Bangladesh. Since marriage between 13-15 years leads to early pregnancy, which can have severe health consequences for both mothers and newborns including malnutrition, morbidity, mortality and motivate disempowerment of girls and women, it is important to address this age group.

The investigators will conduct a cluster-randomized controlled trial in which n=1200 girls age between 13 to 15 years in after-school Adolescent Clubs will participate in a 24-month program teaching women's empowerment through hands-on workshops.

The research will divide participants into two groups: EHFP group and control group.

The EHFP Group will receive Helen Keller's EHFP model-which involves homestead food production, nutrition and WASH education and gender transformative sessions. The control group will not receive the above. Both groups will receive interventions related to parental awareness sessions, community awareness-raising activities, adolescent group sessions involving awareness on the benefit of delayed marriage and empowerment, SRH and basic life-skill trainings. It is hypothesized that the addition of the EHFP program will provide increased production and consumption of nutrient rich foods, increased income of the households through the sale of surplus produce, and increased self-efficacy and decision making by adolescents due to increased knowledge and skills- resulting increased food security and nutrition and ultimately delay of child marriage. A formative research will be conducted in a participatory approach with adolescents and their parents to contextualize the SBC messages and strategies.

Location: The intervention will be placed in Debhata sub-district of Satkhira district in Khulna Division. Since other sub-districts of Satkhira District are already under covered by the Nobo Jatra (the new journey) project implemented by World Vision with the funding support from USAID where the improvement of adolescent nutrition is a major component, investigators decided not to select these sub-districts covered by other similar type of project to avoid any sort of distortion in the trial.

In this cluster randomized controlled trial, blinding will not be possible during study delivery; participants and field staff will know whether a participant is in a control or EHFP cluster. For cluster randomization, 74 Adolescent Clubs (clusters, each Adolescent Club containing approximately 1,110 adolescent participants) will be randomized to one of the two study arms, control or EHFP, using a 1:1 ratio, computer-generated randomization schedule.

Sample size estimation.

The investigators will recruit n=1200 participants (from approximately 80 clusters) in Khulna Division, southern Bangladesh. The intervention will be placed in Debhata sub-district of Satkhira district in Khulna Division. Since other sub-districts of Satkhira District are already under covered by the Nobo Jatra (the new journey) project implemented by World Vision with the funding support from USAID where the improvement of adolescent nutrition is a major component, investigators decided not to select these sub-districts covered by other similar type of project to avoid any sort of distortion in the trial.

The sample has been calculated for a two-level cluster randomized trial, where girls are nested within clusters randomly assigned to each of the three two study arms.

The major impact variables considered to determine the sample size estimation are anemia status, dietary diversity and prevalence of child marriage of the adolescents. The villages in each arm are expected to be comparable and geographically separated to avoid contamination. The investigators will set the power at 80%, alpha at 5% and assume the cluster size (c) equal to 15. With an intra-class correlation of 0.05, the required number of clusters is 74. Thus, investigators will create 74 clusters in total, with 37 clusters with a total of 555 girls aged 13 to 15 years per study arm. Overall, the intervention will target to reach 1,110 adolescent girls in the 2 intervention arms over the 24 months intervention. To ensure enough number of clusters and sample, investigators decided to go beyond the minimum number of both cluster and sample (74 clusters and 1110 samples) for this study. Thus, for both EHFP and control group, the investigators considered 40 cluster totaling 600 samples (40 X 15) for each arm.

Training: All data collection staff will be rigorously trained on survey methodology. This training will cover all topics required for the implementation of the data collection, including locating/ selecting of respondent households and obtaining consent. All training modules include both theory and practical exercises. Model adolescents will be hired for classroom practice so that the data collectors will be familiar with the questionnaire and anthropometric measurements in order to collect data using appropriate techniques. The training will include questionnaire pre-testing to practice data collection and to find any issues with the survey instrument. A major focus of training will be ensuring that the field workers learn to minimize bias when performing interviews and recording data. Three separate batches of trainings will be organized for; a) household questionnaire b) anthropometry measurements.

Data management and analysis: Participants will be given a unique alpha-numeric study ID code. This unique identifier will not be derived from personal identifiers. A key linking the subject code to participant information will be kept on a password-protected computer in a secure area in the Helen Keller International (HKI) office in Dhaka, Bangladesh. There is no need for co-investigators elsewhere to have information linking participant names with their unique identifier.

All electronic data files will be stored on password-protected computers and/or secure servers accessible only to members of the research team. Archived electronic data files and any hard copies of data (consent forms) will be stored in locked filing cabinets in locked research rooms at HKI Bangladesh. Once all data is collected, all information will be de-identified. Only the study Principal Investigator will have access to the master list once data collection is complete; otherwise, all data will be completely de-identified.

All paper copies of consent forms and questionnaires will be retained for at least 5 years after publication of results. All data will be stored on an external hard-drive, in a locked drawer, in the Principal Investigator's locked office for a minimum of 25 years. After this time, all paper copies of consent forms will be shredded, and the hard drive deleted and physically destroyed.

All data will be entered into STATA/SPSS for analysis. Descriptive statistics will be computed for all variables: mean (SD) for continuous variables (age, monthly household income), or n (%) for categorical variables (education level). The investigators will compare the control and EHFP groups using independent t-tests or x2 tests.

Utilization of Results: It is expected that the findings of this study will contribute to the important discourse of empowering and supporting adolescents to prevent child marriage and improve food security and nutrition outcomes, as well as informing future programming for HKI program in Bangladesh and other countries in Asia and Africa and development partners, while at the same time providing evidence-based advocacy for national nutrition and livelihoods strategies and programs. Findings from this project will improve the awareness and understanding among policymakers, think tanks, development community and general public in developing countries including Bangladesh about the efficacy of a gender-transformative EHFP program to prevent child marriage. Based on the critical findings, the project will not only develop new policy but will also shaping the existing policies through identifying the gaps and appropriate context.

ELIGIBILITY:
Inclusion Criteria:

* Not be married,
* Are not sick
* Have never been pregnant,
* Be aged 13-15 years,
* Be willing to attend monthly workshops at their local Adolescent Club,
* Provide written assent to participate from adolescent, and have their primary caregiver (e.g. father/mother) provide written consent for participation,
* Have access to a minimum of about 60 sq.m (1.5 decimal) of homestead land available for EHFP activities at their home.

Exclusion Criteria:

* Not ill or in unhealthy condition

Ages: 13 Years to 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Adolescent girls age between 13 to 15 years
Enrollment: 1200 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2023-03-15 (Estimated)

PRIMARY OUTCOMES:
Prevalence of child marriage | Baseline to twenty four months of the intervention
  This is a continuous variable and the goal is to delay the marriage of the adolescent girl until after 16th birthday.
Adolescent nutrition status-Anemia | Baseline to twenty four months of the intervention
  Anemia will be measured by hemoglobin concentration in the blood and, for this particular indicator, will be collected among adolescent girls (13-15 years). Non-pregnant adolescent girls with a hemoglobin concentration less than 12g/dl will be classified as anemic. The numerator for this indicator is the sample-weighted number of anemic adolescent girls 13-15 years in the sample. The denominator is the sample-weighted number of adolescent girls 13-15 years in the sample with hemoglobin data.
Household income | Baseline to twenty four months of the intervention
  Monthly household income will be measured in US$ by observing changes from baseline to endline
Adolescent nutrition status-Underweight | Baseline to twenty four months of the intervention
  BMI is an anthropometric index of weight and height that is defined as body weight in kilograms divided by height in meters squared. BMI is used to assess underweight status of adult and adolescents.

SECONDARY OUTCOMES:
Food security status of the household | Through study completion, an average of 4 months
  The HFIAS score is a continuous measure of the degree of food insecurity (access) in the household in the past four weeks (30 days). First, a HFIAS score variable will be calculated for each household by summing the codes for each frequency-of-occurrence question out of the nine set of questions. Before summing the frequency-of-occurrence codes, the data analyst will code frequency-of-occurrence as 0 for all cases where the answer to the corresponding occurrence question was "no". If the respondent answered "yes" to an occurrence question, a follow-up question will be asked to determine whether the condition occurred rarely (once or twice), sometimes (three to ten times) or often (more than ten times) in the past four weeks. The maximum score for a household will be 27 (if the household response to all nine frequency-of-occurrence questions was "often", coded with response code of 3); the minimum score will be 0 (the household responded "no" to all occurrence questions) The higher the
Adolescent empowerment and participation in household decision-making | Through study completion, an average of 4 months
  Adolescents' self efficacy will be assessed using the General Self Efficacy (GSE) scale correlated to emotion, optimism, work satisfaction; negative coefficients will be used measure depression, stress, health complaints, burnout, and anxiety using this same measure
Adolescent nutrition status-Dietary diversity | Through study completion, an average of 4 months
  Minimum Dietary Diversity - Women (MDD-W) captures the proportion of women of reproductive age in the FFP project implementation areas who are consuming a minimum dietary diversity. A woman of reproductive age will be considered to consume a minimum dietary diversity if she consumes at least five of 10 specific food groups in the previous 24 hours. MDD-W uses 10 food groups, while WDDS uses nine.

CONTACTS AND LOCATIONS:
Overall Officials: Aminuzzaman Talukder, MPH, Principal Investigator — Helen Keller International
Locations (1):
- Helen Keller International, Sātkhira, Khulna Division, Bangladesh

REFERENCES:
- [Background] Helen Keller International (HKI), James P Grant School of Public Health (JPGSPH). State of Food Security and Nutrition in Bangladesh: 2013. Dhaka; 2014.
- [Background] BDHS. Bangladesh Demographic and Health Survey 2014. 2014. 1-354 p.
- [Background] Ainul S, Bajrachrya A, Reichenbach L. Adolescents in Bangladesh: A Situation Analysis of Programmatic Approaches to Sexual and Reproductive Health Education and Services. Popul Counc Evid Proj. 2017;(January):62.
- [Background] NIPORT. Bangladesh Demographic Health Survey 2007. Natl Inst Popul Res Train. 2007;1-381.
- [Background] NIPORT. Bangladesh Demographic and Health Survey 2014. Dhaka, Bangladesh, and Rockville, Maryland, USA. 2015.
- [Background] Dixon-Mueller R. How young is "too young"? Comparative perspectives on adolescent sexual, marital, and reproductive transitions. Stud Fam Plann. 2008 Dec;39(4):247-62. doi: 10.1111/j.1728-4465.2008.00173.x. PMID 19248713
- [Background] Dick B, Ferguson BJ. Health for the world's adolescents: a second chance in the second decade. J Adolesc Health. 2015 Jan;56(1):3-6. doi: 10.1016/j.jadohealth.2014.10.260. PMID 25530601
- [Background] MoWCA. কিশোর-কিশোরী ক্লাব - Adolescent Program of Bangladesh [Internet]. 2017. Available from: https://mowca.gov.bd/site/notices/f64412aa-e606-47ae-ab7c-63848d74f8ec/Kishore-Kishori-club-project-review-meeting
- [Background] Amin S, Ahmed J, Saha J, Eashita H, Haque F. Delaying child marriage through community-based skills-development programs for girls: Results from a randomized controlled study in rural Bangladesh.
- [Background] Coates J, Swindale A, Bilinsky P. Household Food Insecurity Access Scale (HFIAS) for Measurement of Food Access: Indicator Guide. Washington, D.C.; 2007.
- [Background] FANTA, FAO. Introducing the Minimum Dietary Diversity - Women (MDD-W) Global Dietary Diversity Indicator for Women. 2014;2014-5. Available from: http://www.fantaproject.org/monitoring-and-evaluation/minimum-dietary-diversity-women-indicator-mddw
- [Background] World Food Programme. Food consumption analysis: Calculation and use of the food consumption score in food security analysis [Internet]. Rome, Italy; 2008. Available from: http://library1.nida.ac.th/termpaper6/sd/2554/19755.pdf
- [Background] Home - Equity Tool [Internet]. [cited 2021 Jan 3]. Available from: https://www.equitytool.org/
- [Background] Schwarzer, R., & Jerusalem M (1995). General Self-Efficacy Scale (GSE). 1995.
- [Background] Bangladesh Multiple Indicator Cluster Survey 2012-2013. Progotir Pathey: Final Report. Dhaka, Bangladesh.: Bangladesh Bureau of Statistics (BBS) and UNICEF Bangladesh.; 2013.
- [Background] HKI. State of food security and nutrition in Bangladesh: 2013. 2014
- [Background] Human Rights Watch. Marry Before Your House is Swept Away. 2015.
- [Background] JPGSPH. The state of the world's children. 2016. 1-63 p.
- [Background] NIPORT. BANGLADESH DEMOGRAPHIC AND HEALTH SURVEY 2016. 2016.
- [Background] Karim N, Greene M, Picard M. The cultural context of child marriage in Nepal and Bangladesh: findings from CARE's tipping point project community participatory analysis: research report. 2016
- [Background] Bangladesh Bureau of Statistics and UNICEF Bangladesh. A Scoping Analysis of Budget Allocations for Ending Child Marriage in Bangladesh 2017. 2018.
- [Background] ICRW, Plan. Asia Child Marriage Initiative : Summary of Research in Bangladesh, India and Nepal. UNICEF Glob database. 2013
- See also: Adolescent Program of Bangladesh [Internet]. 2017 — https://mowca.gov.bd/site/notices/f64412aa-e606-47ae-ab7c-63848d74f8ec/Kishore-Kishori-club-project-review-meeting
- See also: Home - Equity Tool [Internet]. [cited 2021 Jan 3]. Available — https://www.equitytool.org/
- See also: World Food Programme. Food consumption analysis: Calculation and use of the food consumption score in food security analysis [Internet]. Rome, Italy; 2008. — http://library1.nida.ac.th/termpaper6/sd/2554/19755.pdf